CLINICAL TRIAL: NCT03795987
Title: TNT/NW: Traumatic Nightmares Treated by NightWare (To Arouse Not Awaken)
Brief Title: Traumatic Nightmares Treated by NightWare (To Arouse Not Awaken)
Acronym: TNT/NW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NightWare (Industry)
Collaborators: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NW101001
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Stress Disorders, Post-Traumatic; Combat Disorders; Ptsd; Nightmare; Nightmares, REM-Sleep Type; Nightmare Disorder With Associated Non-Sleep Disorder
Keywords: PTSD; Nightmare; Nightmare Disorder; Post-traumatic stress disorder; Veteran; Digital therapeutic; Digital medicine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Open Label Treatment Arm (Experimental): Intervention with NightWare Therapeutic System
  Interventions: Device: NightWare Therapeutic System

INTERVENTIONS:
Device: NightWare Therapeutic System — A wearable digital therapeutic system that will measure physiologic data when worn during sleep to deliver a mild vibration via the watch to elicit arousal thereby disrupting nightmares. This detection and stimulation sequence will be performed according to NightWare's proprietary algorithm.

SUMMARY:
This study will provide preliminary estimates of safety and efficacy of the NightWare digital therapeutic system (iPhone + Apple watch + proprietary application) for the treatment of nightmare disorder associated with post-traumatic stress disorder (PTSD)-related sleep disturbance and the impact of improved sleep with the NightWare digital therapeutic system. The investigators hypothesize that the NightWare digital therapeutic system will significantly improve sleep quality in participants with PTSD-Related nightmares and poor sleep quality.

DETAILED DESCRIPTION:
Nightmares are a common problem affecting 2-8% of the general population and a higher proportion of clinical populations. The negative consequences of untreated nightmares are significant and include impaired quality of life, sleep deprivation (often resulting in an increased intensity of nightmares), insomnia, daytime sleepiness, and fatigue. Untreated nightmares can also exacerbate the symptoms of underlying psychological dysfunction in people with depression and anxiety, leading to poor occupational and or social functioning. Nightmares can be idiopathic or associated with the use (or withdrawal) of certain medications or substances, or associated with disorders including PTSD.

NightWare (Minneapolis, MN) has developed a novel approach to the treatment of nightmares. Through the use of a smartwatch-based application that senses physiologic parameters, the participant is aroused from sleep (without awakening the participant) so that the nightmare is interrupted prior to reaching a threshold of severity in which the participant would awaken in distress. Seconds later the participant returns to sleep without having experienced a nightmare. This approach avoids risk from pharmacological treatment, avoids exacerbation of symptoms from image rehearsal therapy and allows for a simple method with easily achieved adherence compared to existing treatments.

The NightWare digital therapeutic system consists of a proprietary software application installed on a smartwatch. The application has been effective in focus groups when used on both Apple smartwatches and Motorola smartwatches. For the purposes of this study, the investigators will be using only the Apple (Cupertino, CA) 3rd generation smartwatch and the Apple iPhone. The NightWare application uses physiological markers obtained via the smartwatch to determine by proprietary algorithm whether a participant is in the early stages of a nightmare, but has not yet awoken in distress. As directed by the algorithm, the smartwatch then applies varying degrees of vibratory stimulation to the wrist over variable lengths of time with the intention of arousing the participant from sleep without eliciting an awakening.

ELIGIBILITY:
Inclusion Criteria:

* Veteran Enrolled in the Minneapolis/St. Cloud VAHCS.
* Diagnosis of PTSD via American Psychiatric Association PTSD diagnostic criteria in the fifth edition of its Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
* Equal to or older than 22 years of age.
* Proficient in both reading and writing in the English language.
* Pittsburgh Sleep Quality Index (PSQI) score 10 or higher.
* Epworth Sleepiness Scale (ESS): On question #8 any score above "0" will prompt an additional question: Do you drive ("get behind the wheel") when you are drowsy? The answer must be "No" to be enrolled in the study due to safety concerns.
* Have repetitive nightmares contributing to disrupted sleep as reported by the patient
* Wireless Internet and two power outlets where they sleep
* Prazosin use; if yes, the patient may be included if tapered by prescribing provider. Taper must be completed and subject must be off prazosin for 2 days prior to enrollment.

Exclusion Criteria:

* Patient Health Questionnaire-9 (PHQ-9) score greater than or equal to 20. A score of 1 or more on the suicide ideation item of the PHQ-9 will trigger a risk assessment.
* Uncontrolled atrial fibrillation
* Current use of varenicline
* Current use of beta-blockers (unless ophthalmic solutions)
* Current use of non-dihydropyridines
* Current use of Prazosin for the treatment of nightmares (can include patients 2 days following taper and discontinuation) This would be coordinated with the prescribing provider
* Circadian rhythm disruption on a regular basis (shift-work)
* Known diagnosis of Obstructive Sleep Apnea
* Diagnosis of an active disorder of arousal from non-rapid eye movement sleep
* Diagnosis of rapid eye movement sleep behavior disorder
* Diagnosis of narcolepsy
* Alcohol Use Disorders Inventory Test (AUDIT) (score of 8 or higher)
* Drug Abuse Screening Test-10 (DAST-10) (score greater than 2)
* Suspicion of nightmares being secondary to substance abuse or withdrawal
* Diagnosis or suspicion of dementia
* Previous or foreseeable legal proceedings involving nightmares or trauma
* Nocturia that causes awakening from sleep
* Known sleepwalking
* Acting out of dreams prior to PTSD trauma

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Change in global score on the Pittsburgh Sleep Quality Index (PSQI) from Day 0 to Day 60 | 0-60 days
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality. This outcome is the difference between the global score on the Pittsburgh Sleep Quality Index (PSQI) score at baseline (Day 0) and average global PSQI score across the four post-treatment initiation assessments (Days 14, 30, 44 and 60).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Karlin, MD MA, Study Chair — NightWare
Locations (1):
- Minneapolis VA Healthcare System, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No